CLINICAL TRIAL: NCT06583473
Title: The Effectiveness of Integrated Interactive Digital Health Application and Telemonitoring in Patients with Heart Failure and Reduced Ejection Fraction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hsiao Fu-Chih (Other)
Responsible Party: Sponsor-Investigator, Hsiao Fu-Chih, Doctor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HFApp
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Health Behavior
Keywords: Heart Failure; Interactive digital health application
MeSH Terms: conditions — Heart Failure; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interactive digital health care (Experimental): The "Intelligent Interactive Personal Management System for Heart Failure" and Bluetooth-enabled devices for remote monitoring of blood pressure and weight.
  Interventions: Behavioral: Interactive digital health application
- Standard care (No Intervention): The control group will continue to receive standard medical care.

INTERVENTIONS:
Behavioral: Interactive digital health application — The study program will provide an integrated interactive digital health application (LINE app on smartphones, incorporating information about biodata recording, health education, questionnaires, and online Q&A)
  Arms: Interactive digital health care

SUMMARY:
Patient Source: Patients discharged from the cardiology ward with heart failure.

Intervention Group: Prior to discharge, patients will be provided with and instructed on how to use the "Intelligent Interactive Personal Management System for Heart Failure" as well as a "Bluetooth-enabled blood pressure monitor and scale for remote data transmission."

Control Group: Patients will receive standard medical care.

Assessment Method: The Health-Related Quality of Life Questionnaire (EQ-5D), Kansas City Cardiomyopathy Questionnaire (KCCQ-12), and Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being; The 12-item Spiritual Well-Being Scale (FACIT-Sp-12) will be completed before discharge, and at 1 month, 6 months, and 12 months post-discharge. The average time to complete the questionnaires is 10-15 minutes. Additionally, cardiovascular events and readmission rates will be tracked and analyzed over a 1-year period.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with heart failure

Exclusion Criteria:

Inability to independently stand or get out of bed. Unstable condition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Heart failure re-hospitalization rate | 1 Year
  The rate of heart failure re-hospitalization
Kansas City Cardiomyopathy Questionnaire | 1 Year
  The KCCQ-12 is a validated health status measure for patients with HF. It contains four subdomains: Physical Limitation, Symptom Frequency, Quality of Life, and Social Limitations. Each subdomain provides an individual score from 0 to 100, with 0 denoting the worst and 100 the best possible health status. The mean of the four subdomain scores are presented as a summary score, with differences of 5 points or greater considered to be clinically important.
EQ-5D | 1 Year
  The EQ-5D-5L is a widely used health status measure with two parts. The first part evaluates health across five dimensions: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN/DISCOMFORT, and ANXIETY/DEPRESSION, each with five response levels. This generates a health state profile, which can be assigned a summary index score based on societal preference weights, or "utilities," for calculating QALYs in health economics. Scores range from less than 0 (death or worse) to 1 (full health), with higher scores indicating better health utility. The second part of the questionnaire is a visual analogue scale (VAS) where patients rate their perceived health from 0 (worst imaginable health) to 100 (best imaginable health).
FACIT-Sp-12 | 1 Year
  The Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT-Sp-12) is a 12-item scale designed to measure spiritual well-being in individuals with chronic illnesses. Possible scores range from 0 to 48, with higher scores reflecting greater spiritual wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No
In the early phase after the diagnosis of HFrEF, self-monitoring of the blood pressure, pulse rate, and body weight at home, enhancement of the knowledge and self-awareness of the disease, and regular outpatient follow-up and health education are key elements in improving adherence to pharmacotherapies; and improving quality of holistic health care, including physiological, psychological, and social aspects.